CLINICAL TRIAL: NCT04926909
Title: The Relationship Between Serum Cystatin C and PET-DAT Study in Patients With Parkinson's Disease
Brief Title: Study on Serum Cystatin C and PET-DAT in Patients With Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-079
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-03

CONDITIONS: Parkinson's Disease
Keywords: Cystatin C, PET-DAT
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month

SUMMARY:
To investigate the relationship between serum cystatin C and dopamine receptor(DAT) loss in patients with parkinson's disease(PD)

DETAILED DESCRIPTION:
Number of people suffered from Parkinson disease (PD) is increasing every year. PET imaging of dopamine transport receptors（DAT） serves as the gold standard for the diagnosis and monitoring of PD development. However, due to high costs and radiation reasons, it is not suitable for long-term follow-up. Serum cystatin C can be easily obtained and cheap as an indicator. In recent years, studies have gradually found that it is related to the progression of H&Y staging of Parkinson's disease. To this extent, we want to further explore whether it can reflect the loss of DAT in the brain. Explore whether it can partially replace the role of DAT imaging for future clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 80 years and whose laboratory results included the levels of serum Cystatin C within a month from the PET-DAT were recruited.

Exclusion Criteria:

* To make the study cohort more homogeneous, PD patients with either a long-standing duration (≥5 years) or advanced Hoehn and Yahr (H&Y) staging (≥3) were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pearson correlation analysis is planned, and the sample size is calculated with PASS 15.0 software. 121 participants required after sample size calculation. The calculation parameters are as follows: Power = 0.90, α=0.05, ρ0 = 0.0, and ρ1 = 0.3.
Sampling Method: Probability Sample
Enrollment: 121 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Cystatin C assesses the loss of dopaminergic neurons | through study completion, an average of 1 year
  Explore whether Cystatin C can respond to the loss of dopaminergic neurons

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China